CLINICAL TRIAL: NCT04412213
Title: Correlation of Family History, Age at Onset and Severity of Stuttering in School-age Children
Brief Title: Correlation of Family History, Age at Onset & Severity of Stuttering
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherine Khaled Mohammed Elderwy, Resident of Phoniatrics at Assiut Psychiatric Health Hospital, Assiut University
Other Study IDs: family history of stuttering
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Stuttering, Childhood
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children of possitive family history of stuttering
  Interventions: Other: Stuttering severity instrument for school-age children (SSI-3 Arabic version)
- children of negative family history of stuttering
  Interventions: Other: Stuttering severity instrument for school-age children (SSI-3 Arabic version)

INTERVENTIONS:
Other: Stuttering severity instrument for school-age children (SSI-3 Arabic version) — Stuttering severity instrument for school-age children (SSI-3 Arabic version) for measuring stuttering severity Stanford Binet test version 4 to evaluate the mentality (IQ)
  Other Names: Stanford Binet test version 4

SUMMARY:
The aim of this study is to Detect the influence of the family history of stuttering (distance of relative) on the onset and severity of stuttering in children in these families. Also to explore developmental differences among young stutterers.

ELIGIBILITY:
Inclusion Criteria:

* 1-Age: from 7 to 15 years old. 2-Gender: both sexes will be included in the study. 3-The participants are diagnosed as stutterers by an expert phoniatrician. 4-Children will be accepted only if full information is provided concerning the presence or absence of family history of stuttering, from both paternal and maternal sides of the family, and the age of onset of stuttering manifestations. 5-Mentality: IQ is 80 or more

Exclusion Criteria:

* 1-Age below 7 years or above 15 years. 2-Failure to provide full information concerning the presence or absence of family history of stuttering, from both paternal and maternal sides of the family, or age of onset of stuttering manifestations.. 3- IQ less than 80

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 50 stuttering childern, age between 7 and 15 years, with an IQ =80 or more
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
assess the correlation between family history, age of onset and severity of stuttering | year
  family history may affect the onset of stuttering and its severity. children with possitive family history of stuttering may develope stuttering earlier than children with negative family history and stuttering could be more severe in the first group.

REFERENCES:
- [Background] Yairi E, Ambrose N. Onset of stuttering in preschool children: selected factors. J Speech Hear Res. 1992 Aug;35(4):782-8. doi: 10.1044/jshr.3504.782. PMID 1405533
- [Background] Buck SM, Lees R, Cook F. The influence of family history of stuttering on the onset of stuttering in young children. Folia Phoniatr Logop. 2002 May-Jun;54(3):117-24. doi: 10.1159/000063407. PMID 12077503